CLINICAL TRIAL: NCT05123456
Title: Risk of Osteoarthritis of the Knee at Least 5 Years After ACL Reconstruction: Comparative Study Between an Isolated ACL Reconstruction and a Reconstruction Combining ACL and ALL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other); Private Hospital Jean Mermoz (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2018-A02447-48
Record Dates: First submitted 2021-11-09; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: ACL; Anterior Curciate Ligament; Anterolateral Ligament; Knee Injuries; ALL
MeSH Terms: conditions — Knee Injuries | interventions — X-Rays

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient operated with isolated ACL knee reconstruction (Experimental)
  Interventions: Procedure: Radiography
- Patient operated with ACL and ALL knee reconstruction (Experimental)
  Interventions: Procedure: Radiography

INTERVENTIONS:
Procedure: Radiography — Comparative X-ray of the single knee at 30 ° flexion.

SUMMARY:
The main objective of this study is to compare, with a minimum follow-up of 5 years, the prevalence of femoro-tibial osteoarthritis after an isolated ACL ligamentoplasty or after an ACL ligamentoplasty combining ACL and ALL.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent an isolated Anterior Cruciate Ligament (ACL) reconstruction or a combined ACL and anterolateral ligament reconstruction (Extra Articular Plasty) between January 1, 2011 and March 31, 2012.
* Patients affiliated or beneficiaries of a social security scheme
* Patients who have given their express consent.

Exclusion Criteria:

* Patients with pediatric ACL reconstruction technique
* Patients with a complex associated gesture such as osteotomy or ligamentoplasty other than extra articular plastic surgery.
* Contraindication to a radio control (pregnancy)
* Patient's refusal to participate in the study
* Protected patients: Adults under guardianship, curatorship or other legal protection, deprived of their liberty by judicial or administrative decision; Pregnant, breastfeeding or parturient woman; Hospitalized without consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of the prevalence of femoro-tibial osteoarthritis | 1 day
  The prevalence of femoro-tibial osteoarthritis will be assessed by the percentage of patients with cartilage damage to the femoro-tibial compartments on a single X-ray of the face compared to 30 °of flexion.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital privé Jean Mermoz, Lyon, France

REFERENCES:
- [Derived] Shatrov J, Freychet B, Hopper GP, Coulin B, El Helou A, An JS, Vieira TD, Sonnery-Cottet B. Radiographic Incidence of Knee Osteoarthritis After Isolated ACL Reconstruction Versus Combined ACL and ALL Reconstruction: A Prospective Matched Study From the SANTI Study Group. Am J Sports Med. 2023 Jun;51(7):1686-1697. doi: 10.1177/03635465231168899. Epub 2023 May 8. PMID 37154412